CLINICAL TRIAL: NCT04415060
Title: SedAting With Volatile Anesthetics Critically Ill COVID-19 Patients in ICU: Effects On Ventilatory Parameters And Survival. Multicentre Open-label, Pragmatic, Randomized Controlled Trial and a Parallel Prospective (Non-randomized) Cohort Study
Brief Title: SedAting With Volatile Anesthetics Critically Ill COVID-19 Patients in ICU: Effects On Ventilatory Parameters And Survival
Acronym: SAVE-ICU
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2149
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-07

CONDITIONS: Covid19; Hypoxic Respiratory Failure
Keywords: sedation; ICU; volatile anesthetics
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Multicentre open-label, pragmatic, randomized controlled trial and a parallel prospective (non-randomized) cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inhaled - volatile anesthetic (Experimental): The ICU patient will be randomized to either Isoflurane or Sevoflurane, whichever is available at the hospital. Dosage will be modified as per health care team guidance for the best treatment of the participant.
  Interventions: Drug: Isoflurane Inhalant Product; Drug: Sevoflurane inhalant product
- Standard Care (No Intervention): The ICU patient will be randomized to standard of care, which is any IV sedation supplied by the hospital. Dosage will be modified as per health care team guidance for the best treatment of the participant.
- Non-randomized (No Intervention): In this arm, ICU patients who cannot be randomized will receive inhaled or IV sedation as per available in their unit. This is done to try to obtain the maximum amount of information available from the patients present to our ICUs.

INTERVENTIONS:
Drug: Isoflurane Inhalant Product — Isoflurane will be administered using an inhalation device
  Arms: Inhaled - volatile anesthetic
Drug: Sevoflurane inhalant product — Sevoflurane will be administered using an inhalation device
  Arms: Inhaled - volatile anesthetic

SUMMARY:
Patients suffering lung failure, possibly from COVID-19 or hypoxic lung failure, will need life-saving support from a breathing machine. Any patient needing this support requires drugs to keep them sleepy, or "sedated" to be comfortable on this machine. Sedation is made possible by using drugs given through a vein. Unfortunately, these drugs are in short supply worldwide due to the high number of COVID-19 patients needing these machines.

Another way to provide sleep is by using gases that are breathed in. These are used every day in operating rooms to perform surgery. These gases, also called "inhaled agents" can also be used in intensive care units and may have several important benefits for patients and the hospital. Research shows they may reduce swelling in the lung and increase oxygen levels, which allows patients to recover faster and reduce the time spent on a breathing machine. In turn, this allows the breathing machine to be used again for the next sick patient. These drugs may also increase the number of patients who live through their illness. Inhaled agents are widely available and their use could dramatically lesson the pressure on limited drug supplies.

This research is a study being carried out in a number of hospitals that will compare how well patients recover from these illnesses depending on which type of sedation drug they receive. The plan is to evaluate the number who survive, their time spent on a breathing machine and time in the hospital. This study may show immediate benefits and may provide a cost effective and practical solution to the current challenges caring for patients and the hospital space, equipment and drugs to the greatest benefit. Furthermore, the study will be investigating inflammatory profile and neuro-cognitive profiles in ventilated patients. Finally, this trial will be a team of experts in sedation drugs who care for patients with proven or suspected COVID-19 who need lifesaving treatments.

DETAILED DESCRIPTION:
Multicentre open-label, pragmatic, randomized controlled trial and a parallel prospective (non-randomized) cohort study conducted in ICUs and ICU enabled environments caring in critically ill COVID-19 and non-COVID hypoxic respiratory failure patients.

Participants will be mechanically ventilated and will be variably randomized, within 72 hours of start of sedation treatment, in a 1:1 ratio to either an intravenous or inhaled volatile-based sedation arm depending on availability of sedative drugs for both arms. Stratification will be done by:

1. Age ≥ 65 years
2. participating centre
3. PaO2/FiO2 ratio of 150

Patients who cannot be randomized (due to technical or resource issues in some areas of the hospital) will be entered into the parallel prospective (non-randomized) cohort study and will receive intravenous or inhaled sedation as able in their designated unit.

Sedation will be administered according to standard sedation practice and in keeping with current guidelines.

Participants will be followed:

* daily in ICU until 30 days after enrollment, ICU discharge or death, whichever occurs first;
* at 30 days after last dose of drug administration by telephone or through the hospital healthcare database;
* at 60 days, 90 days, and 365 days after enrollment by telephone and/or through data linkages with a provincial or hospital or state healthcare database;
* Participants will have the option to participate in the neuro-cognitive and / or biomarker assessments

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Mechanically ventilated and expected to remain mechanically ventilated at the end of the next day
3. Receiving IV sedation by infusion or bolus for ≤72 hours to facilitate mechanical ventilation Transferred patients with escalating ventilation needs are eligible for recruitment within ≤72 hours of sedation commenced within the participating trial site that they were transferred to.

   Note: Intravenous sedation required to support mechanical ventilation includes use of one or more of the following agents: benzodiazepines, propofol, ketamine, barbiturates, alpha-2 agonist, opioids. Patients receiving intravenous opioids only i.e., fentanyl ≥ 50mcg/hour, hydromorphone ≥ 0.4mg/hour (or bolus q1h) for analgesia and sedation or agitation to assist mechanical ventilation are eligible for inclusion.
4. Mechanically ventilated patients +/- extracorporeal membrane oxygenation (extracorporeal life) support with:

   1. Proven or suspected (under investigation) COVID-19, or
   2. COVID-19 negative patients who have a PaO2FiO2 ratio ≤300 measured with arterial blood gas at least once during the 12 hours prior to enrollment.

Note: If arterial blood gas measurement is unavailable, the PaO2 can be imputed from the pulse oximetry measurement

Exclusion Criteria:

1. Contraindications to sedatives, such as propofol infusion syndrome or malignant hyperthermia;
2. Known allergy to any of the ingredients or components of the investigational products; sevoflurane or isoflurane;
3. Suspect or evidence of high intracranial pressure;
4. Severe brain injury that is likely to lead to sustained very low conscious levels or vegetative state
5. Severe neuromuscular disorder for example amyotrophic lateral sclerosis, Gullian Barre Syndrome that are the primary cause of needing ICU admission and mechanical ventilation
6. One-lung ventilation or pneumonectomy;
7. Ideal estimated tidal volume too low for delivery of inhaled agents. Target (6ml/kg) < 200ml;
8. Use of inhaled prostacyclin which is contraindicated in the presence of a miniature vaporizer (i.e., Anesthesia Conserving Device). This agent has a high viscosity that leads to poor vaporization of the volatile agent. Note: Other inhaled pulmonary vasodilators such as nitric oxide can be safely administered in the presence of miniature vaporizers. Use of prostacyclin is permissible with an anesthesia machine and MADM;
9. Known pregnancy
10. Moribund patient not expected to survive >12 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Hospital Mortality | 365 days
  Does the use of inhaled volatile anesthetic-based sedation regimen improve participant hospital mortality as compared to standard intravenous sedation regimen with a 10% difference between groups for 758 participants.

SECONDARY OUTCOMES:
Ventilator-Free Days | 30 days
  Does the use of inhaled volatile anesthetic-based sedation regimen improve participant ventilation outcomes after 30 days post enrollment, as compared to standard intravenous sedation regimen for 200 participants
ICU-Free Days | 30 days
  Does the use of inhaled volatile anesthetic-based sedation regimen improve participant time spent in ICU, 30 days post enrollment, as compared to standard intravenous sedation regimen for 128 participants
Participant Quality of Life at 3 months after discharge | 90 days
  Does the use of inhaled volatile anesthetic-based sedation regimen improve participant quality of life outcomes at 3 months post discharge as compared to standard intravenous sedation regimen for 144 participants. To evaluate the quality of life, the EuroQol-5 Dimensional (EQ5D) survey will be completed at 90 days.
Delirium and Coma Free Days | 14 days
  To evaluate the days alive and free from delirium and coma while in ICU for 14 days after enrollment
Median Daily Oxygenation | 3 days
  To evaluate participant median daily oxygenation (PaO2/FiO2) at 3 days post enrollment
Adjunctive ARDS therapies | 30 days
  To evaluate participant need for adjunctive ARDS therapies (prone, nitric oxide, paralysis, ECMO) during ICU stay
Hospital-Free Days | 60 days
  To evaluate the number of hospital-free days for participants, 60 days after enrollment
Disability | 365 days
  To evaluate participant disability at 3 and 12 months post discharge. The World Health Organization Disabiltity Assessment Score (WHODAS 2.0) will be completed at both timepoints. The scores assigned to each of the items - "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4) - are summed. This method is referred to as simple scoring because the scores from each of the items are simply added up without recoding or collapsing of response categories; thus, there is no weighting of individual items.

CONTACTS AND LOCATIONS:
Locations (13):
- Canada (13):
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - London Health Sciences Centre - University Hospital, London, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hopsital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Centre - Royal Victoria Hospital, Montreal, Quebec
  - Hôpital Sacré-Coeur de Montréal, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec (IUCPQ), Québec, Quebec
  - Universite de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jerath A, Slessarev M, Martin C, D'Aragon F, Carrier FM, Senaratne J, Meggison H, Hooper J, Alexandros Cavayas Y, Goligher EC, Couture EJ, Randall I, Hatzakorzian R, Jacka M, Wiener-Kronish J, Xie Z, Pinto RL, Cuthbertson B; SAVE-ICU Investigators and the Canadian Critical Care Trials Group. Sedating with volatile anaesthetics for COVID-19 and non-COVID-19 acute hypoxaemic respiratory failure patients in ICU (SAVE-ICU): protocol for a randomised clinical trial. BMJ Open. 2025 Oct 13;15(10):e108441. doi: 10.1136/bmjopen-2025-108441. PMID 41083292

DOCUMENTS (1):
  • Statistical Analysis Plan (2026-01-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT04415060/SAP_000.pdf